CLINICAL TRIAL: NCT04065945
Title: Epigenetic Safety of Various Protocols in Assisted Reproductive Technology
Brief Title: Epigenetic Safety of Assisted Reproductive Technology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: International Peace Maternity and Child Health Hospital (Other); Changhai Hospital (Other)
Responsible Party: Principal Investigator, Dan Zhang, Principal Investigator, Women's Hospital School Of Medicine Zhejiang University
Other Study IDs: 2018YFC1005003
Record Dates: First submitted 2019-08-12; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine, granulosa cells, follicular fluid , sperm and semen ,abandoned egg or embryo,villi, decidua, placenta, amniotic fluid, umbilical cord blood, and buccal swabs of the offspring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Couples undergoing ART treatment: Couples in reproductive age undergoing ART treatment in Women's Hospital School of Medicine Zhejiang University, The International Peace Maternity & Child Health Hospital, and Changhai Hospital of Shanghai.
  Interventions: Other: Completion questionnaires/providing biological samples
- Couples getting pregnant naturally: Couples who get pregnant naturally and want to deliver the babies in Women's Hospital School of Medicine Zhejiang University, The International Peace Maternity & Child Health Hospital, and Changhai Hospital of Shanghai.
  Interventions: Other: Completion questionnaires/providing biological samples

INTERVENTIONS:
Other: Completion questionnaires/providing biological samples — Participant completes baseline interview at enrollment, then completes questionnaires and provides biological samples at each scheduled study visit.

SUMMARY:
The primary purpose of the study is to investigate the relationship between different protocols of assisted reproductive technology and the epigenetic safety of the offspring. Different interventions of assisted reproductive technology include controlled ovarian hyperstimulation (COH), in vitro embryo culture, in vitro fertilization(IVF), intracytoplasmic sperm injection(ICSI), frozen-thawed embryo transfer(FET), preimplantation genetic testing(PGT). The investigators are also interested in the relationship between pregnancy outcomes in ART or natural conception and environmental, nutritional and lifestyle factors.

ELIGIBILITY:
Inclusion Criteria:

1. Couples undergoing treatment for infertility or getting pregnant naturally and wanting to deliver their babies in Women's Hospital School of Medicine Zhejiang University, The International Peace Maternity & Child Health Hospital, and Changhai Hospital of Shanghai.
2. Men 22-55 years old
3. Women 20 - 45 years old

Exclusion Criteria:

1. Any individual or couple who is outside of age range .
2. Any couple who don't plan to complete their pregnancy check-up or deliver their babies in Women's Hospital School of Medicine Zhejiang University, The International Peace Maternity & Child Health Hospital, or Changhai Hospital of Shanghai.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study subjects will be recruited from couples seeking treatment of infertility or getting pregnant naturally and wanting to deliver their babies at the Women's Hospital School of Medicine Zhejiang University. Men must be at least 22 years old and women must be at least 20 years to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 1 day after delivery
  Number of women with live births / number of women randomized to the specific group.Live birth is defined as the delivery of any viable infant at 28 weeks or more of gestation after our interventions.
birth weight | 1 day after delivery
  Weight of newborns at delivery.
implantation rate | 11-12 weeks after embryo transfer
  Implantation rate was defined as the percentage of fetal heart beat among total transferred embryos at 12 weeks' gestational age.
clinical pregnancy rate | 6 weeks after embryo transfer
  Clinical pregnancy was defined as an observation of gestational sac via ultrasonography.
congenital anomalies rate | 1 day after delivery
  Congenital anomaly included deformity and development abnormality of any organs or systems.
weight | Change from the date of delivery up to 4 years after delivery
  the weight of offspring
height | Change from the date of delivery up to 4 years after delivery
  the height of offspring
Incidence of mental diseases and metabolic dysfunction | 4 years after delivery

SECONDARY OUTCOMES:
biochemical pregnancy rate | 2 weeks after embryo transfer
  Biochemical pregnancy is defined as numbers of women with an elevated serum β-hCG level of more than 10 mIU/ml.
pregnancy loss rate | 28 gestational weeks in maximum
  Pregnancy loss is defined as any reason that resulted in failure of an embryo to develop, embryonic or fetal death, or spontaneous expulsion of a pregnancy.
ectopic pregnancy rate | 12 gestational weeks in maximum
  Ectopic pregnancy is defined as an embryo implanted outside the uterine.
preterm birth rate | 28 gestational weeks to 37 gestational weeks
  preterm birth is defined as gestational weeks between 28 to 37.
Incidence of moderate to severe ovarian hyperstimulation syndrome(OHSS) | 3 months after controlled ovarian hyperstimulation
  Number of cycles of moderate to severe OHSS/total number of fresh stimulation cycle.
neonatal complication rate | 1 day after delivery
  Neonatal complication includes neonatal respiratory disorders, neonatal cerebral palsy, neonatal encephalopathy and other disease that should been sent into neonatal ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhang, M.D, Ph.D, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided